CLINICAL TRIAL: NCT06629701
Title: A Prospective Randomized Trial of External Vein Graft Support in Surgical Myocardial Revascularization
Acronym: Vest II
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Pilsen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Device Feasibility
Other Study IDs: Vest II
Record Dates: First submitted 2024-10-01; First posted 2024-10-08 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Heart Attack, Revascularization
Keywords: Heart attack, revascularization
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Experimental): Group A will consist of a group of patients who will be sutured with external support for vein grafts.
  Interventions: Device: External support for vein grafts
- Group B (No Intervention): Group B will be without sewn-in external supports.

INTERVENTIONS:
Device: External support for vein grafts — Group A will consist of a group of patients who will be sutured with external support for vein grafts.
  Arms: Group A

SUMMARY:
The aim of the thesis is to compare a group of patients using vein grafts with and without external support, specifically their patency. This is a prospective study with a follow-up plan of 150 patients, in whom the functionality of the grafts will be monitored at time intervals.

DETAILED DESCRIPTION:
One of the most frequently used strategies to restore blood flow in affected coronary arteries in atherosclerotic disease is coronary bypass, or bridging of a narrowed or closed artery and revascularization of the ischemic area of the heart. For coronary artery bypass grafting (CABG), the great saphenous vein (VSM) remains the most commonly used graft, although the longevity of the vein graft is an important limiting factor in monitoring long-term results of CABG. Long-term follow-up found that 25% of vein grafts close within 1 year of surgery, and up to 75% of vein grafts close 10 years after surgery.

External support minimizes pathophysiological processes in the graft. For example, intimal hyperplasia, kinking, graft dilatation or graft suppression and generally improving the hemodynamic flow through the graft should also reduce the formation of thrombus. In this study we follow up the patency and function of vein grafts over a period of 4 years, and compare the resulting data with already available data from other researches.

ELIGIBILITY:
Inclusion Criteria:

* elective cardiosurgical revascularization using VSM vein graft, i.e. patients with MVD findings.

Exclusion Criteria:

* thromboembolic event in the past, long-term warfarinization, mechanical valves, infection during the procedure, urgent procedure, allergy to contrast material, pregnancy, elevated creatinine. A relative contraindication for exclusion from the study is: VSM varicosity, VSM damage during sampling.The age, gender or weight of the patient has no influence on the indication.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Closing of bypass in time | 3 years after the operation
  Primary measures will be closing of the bypass in time, if there will be any.

SECONDARY OUTCOMES:
Chest pain | 3 years after the operation
  Chest pain
Shortness of breath at rest | 3 years after the operation
  Shortness of breath at rest

CONTACTS AND LOCATIONS:
Overall Officials: Viktor Zlocha, MD, Principal Investigator — Head of Cardiac Surgery
Locations (1):
- University Hospital Pilsen, Pilsen, Czech Republic, Czechia

IPD SHARING:
Plan to Share IPD: No